CLINICAL TRIAL: NCT06081075
Title: Newborn Genomics Programme
Status: Recruiting | Type: Observational
Sponsor: Liggins Institute (Other)
Responsible Party: Principal Investigator, Justin O'Sullivan, Professor, Deputy Director, Liggins Institute
Other Study IDs: LIG-2301
Record Dates: First submitted 2023-06-29; First posted 2023-10-12 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Genetic Disease; Newborn Morbidity
MeSH Terms: conditions — Genetic Diseases, Inborn | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Acutely ill neonates with suspected genetic condition, without a clear non-genetic aetiology
  Interventions: Other: Genetic testing

INTERVENTIONS:
Other: Genetic testing — Rapid whole genome sequencing

SUMMARY:
Genomic methods can significantly contribute to all facets of precision medicine, from diagnosis to prevention, therapeutic intervention, and management of acute and chronic illnesses. DNA based methods are already having a considerable impact across healthcare in fields that include: public health, infectious disease monitoring, acute and chronic disease, pharmacogenomics, prenatal testing and diagnosis, and therapeutic development. In this proposal, investigators are focusing on the application of genomic methods in precision medicine - specifically on rapid whole-genome sequencing of parents and children (i.e. a trio) for the identification of diseases that have genetic components.

Goals Primary goal: is to provide safe rapid whole genome sequencing to Neonatal Intensive Care Unit/Pediatric Intensive Care Unit patients.

Secondary goals: 1) Although several groups globally are implementing rapid sequencing of rare disease, these are predominantly in the research space, with many unanswered questions regarding the best way to implement them into a national healthcare system. Each country and their healthcare systems are unique, and valuable knowledge will be gained by implementing this process within a New Zealand context. As part of this the study will measure the impact on the individuals and families.

2) to expand the research team's understanding of non-coding disease-causing variants and methylation changes that contribute to severe disease in early life.

Primary Aims

1. To incorporate long-read RNA sequencing data into the diagnostic rapid Whole Genome Sequencing pipeline to provide a direct measure of the functional outcome of the variants of clinical concern.
2. To measure the clinical utility of analysing non-coding variants in the diagnosis of critically ill children who do not have pathogenic, likely pathogenic, or variants of unknown significance for mendelian disorders.
3. To identify, in a real-world setting within the New Zealand health-care system, the clinical and economic effects of deploying rapid Whole Genome Sequencing-informed rapid precision medicine for critically ill children.

ELIGIBILITY:
Inclusion Criteria:

* Acutely ill inpatient
* Admitted to NICU or PICU between April 2023 - March 2026
* Within 1 week of hospitalization or within 1 week of development of abnormal response to standard therapy for an underlying condition
* Suspected genetic condition, without a clear non-genetic aetiology

Exclusion Criteria:

* Patients whose clinical course is entirely explained by
* Isolated prematurity
* Isolated unconjugated hyperbilirubinemia
* Infection or sepsis with expected response to therapy
* A previously confirmed genetic diagnosis that explains the clinical condition -
* Isolated transient neonatal tachypnoea
* Meconium aspiration syndrome
* Trauma
* Inability to source blood and buccal samples for DNA extraction from at least the mother and child

Ages: 0 Hours to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with suspected genetic conditions, and their families, will be recruited into the study from within the neonatal and paediatric intensive care units (i.e. NICU and PICU, respectively) from around New Zealand
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To incorporate long-read RNA sequencing data into the diagnostic rapid Whole Genome Sequencing pipeline to provide a direct measure of the functional outcome of the variants of clinical concern | June 2025
To measure the clinical utility of analysing non-coding variants in the diagnosis of critically ill children who do not have pathogenic, likely pathogenic, or variants of unknown significance for mendelian disorders. | June 2025
To identify, in a real-world setting within the New Zealand health-care system, the clinical and economic effects of deploying rapid Whole Genome Sequencing-informed rapid precision medicine for critically ill children. | June 2025

CONTACTS AND LOCATIONS:
Locations (1):
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nyaga DM, Tsai P, Gebbie C, Phua HH, Yap P, Le Quesne Stabej P, Farrow S, Rong J, Toldi G, Thorstensen E, Stark Z, Lunke S, Gamet K, Van Dyk J, Greenslade M, O'Sullivan JM. Benchmarking nanopore sequencing and rapid genomics feasibility: validation at a quaternary hospital in New Zealand. NPJ Genom Med. 2024 Nov 8;9(1):57. doi: 10.1038/s41525-024-00445-5. PMID 39516456